CLINICAL TRIAL: NCT05021822
Title: The Effect of Erector Spinae Plane Block on Diaphragma Movement in Laparoscopic Cholecystectomies
Brief Title: The Effect of Erector Spinae Block on Diaphragma Movement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Ülkü Ceren Köksoy, Associate Professor, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-03
Record Dates: First submitted 2021-08-13; First posted 2021-08-26 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Laparoscopic Cholecystectomy; Acute Post-operative Pain; Respiratory Diaphragm
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Block Group (Active Comparator)
  Interventions: Procedure: Erector spinae plane block
- Control Group (No Intervention)

INTERVENTIONS:
Procedure: Erector spinae plane block — Bilateral erector spinae plane block will be performed preoperatively under ultrasound guidance using 15 ml bupivacaine on each side
  Arms: Block Group

SUMMARY:
Laparoscopic cholecystectomy surgeries cause moderate/severe pain and thus can result in shallow breathing, atelectasis and increased opioid consumption in the early postoperative period which in turn cause a longer hospital stay. Erector spinae plane block has been shown to decrease lower thoracic pain after laparoscopic cholecystectomy surgeries. This study aims to investigate the effect of erector spinae plane block on opioid consumption and diaphragma movement after laparoscopic cholecystectomy surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 65
* Patients in American Society of Anesthesiologists Classification I or II
* Elective laparoscopic cholecystectomy surgery performed under general anesthesia

Exclusion Criteria:

* Patient refusal
* Patients who can not provide informed consent or with a known psychiatric disease
* Patients with a known allergy to study drugs
* Patients using anticoagulants and corticosteroids
* Patients with diaphragma hernia, chronic obstructive pulmonary disease, lung cancer
* Patients who are not able to use a patient controlled analgesia device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
Change of Diaphragma excursion | Preoperative measurement-before the erector spina plane block application and postoperative measurement- 30 minutes after extubation
  The change of diaphragma excursion as measured by ultrasound in M-mode from the preoperative period to the postoperative period
Change in Opioid consumption | Postoperative 12 hours: in the first 30 minutes after extubation, 1st hour, 6th hour and 12th hour
  To assess Tramadol consumption measured in mg postoperatively in the first 12 hours after the operation
Change in postoperative pain | Postoperative 12 hours: in the first 30 minutes after extubation, 1st hour, 6th hour and 12th hour
  Postoperative pain will be measured with visual analog scale and numeric scale in the first 12 hours after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ülkü C Köksoy, Ass. Prof., Principal Investigator — Ufuk University Faculty of Medicine Department of Anesthesiology and Reanimation
Locations (1):
- Ufuk Üniversitesi Dr. Rıdvan Ege Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petsas D, Pogiatzi V, Galatidis T, Drogouti M, Sofianou I, Michail A, Chatzis I, Donas G. Erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: a case report. J Pain Res. 2018 Sep 24;11:1983-1990. doi: 10.2147/JPR.S164489. eCollection 2018. PMID 30288093
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392